CLINICAL TRIAL: NCT07070401
Title: The Use of AR / VR in Patients Presenting to the ED With Renal Colic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Community Medical Center, Toms River, NJ (Other)
Responsible Party: Principal Investigator, Greg Neyman, Research Director, Community Medical Center, Toms River, NJ
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-001
Record Dates: First submitted 2025-04-02; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Renal Colic; Kidney Stones, Urolithiasis, Hypocitraturia
Keywords: Renal Colic; Nephrolithiasis; Urolithiasis; Emergency Department; Pain Management; Virtual Reality; Augmented Reality; Audiovisual Stimulation; Patient Anxiety
MeSH Terms: conditions — Renal Colic; Kidney Calculi; Urolithiasis; Nephrolithiasis; Emergencies; Agnosia

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial between Standard of Care vs Standard of Care + Adjunct AR Calming
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Pharmacologic Management (Active Comparator): Patients receive standard of care pharmacologic management at the discretion of the treating provider
  Interventions: Other: Pharmacologic Standard of Care Alone
- AR Adjunct Plus Standard of Care Pharmacologic Management (Experimental): Patients receive adjunct AR Calming App via commercial AR/VR headset in addition to standard of care pharmacologic management at the discretion of the treating provider
  Interventions: Device: Commercial AR/VR Headset with Calming App

INTERVENTIONS:
Device: Commercial AR/VR Headset with Calming App — Commercial AR/VR Headset with Calming App in addition to Pharmacologic Standard of Care
  Arms: AR Adjunct Plus Standard of Care Pharmacologic Management
Other: Pharmacologic Standard of Care Alone — Pharmacologic Standard of Care Alone
  Arms: Standard of Care Pharmacologic Management

SUMMARY:
Utilization of VR / AR Calming as an adjunct to pharmacologic pain management for Renal Colic in Emergency Department Patients

DETAILED DESCRIPTION:
This study will randomize ED patients presenting for presumed renal colic to either standard pharmacologic pain management alone, or pharmacologic management plus use of an adjunct Virtual / Augmented reality calming application using an off-the-shelf VR/AR Headset.

ELIGIBILITY:
Inclusion Criteria:

* Patient self-reported history of nephrolithiasis
* Subjective history suggesting that current presentation is similar to past presentations of nephrolithiasis (character, quality, location, intensity of pain; previous surgical intervention or lithotripsy)
* Patients with self-reported moderate to severe pain on the visual pain scale determined as greater than 5/10
* Normal vital signs (afebrile)
* Agreeable to informed consent as dictated by IRB and local practice
* No contraindications to standard therapy (ie fluids, NSAIDs, opioids, etc.)
* Compliance with the virtual reality treatment
* Keeps the headset on for the duration of the experience
* Understands the instructions

Exclusion Criteria:

* Age < 18 years
* Pregnant
* Individuals with chronic pain conditions such as fibromyalgia (chronic pain may confound results, as patients may have higher than baseline pain levels affecting their response to medications)
* Individuals with severe anxiety or claustrophobia
* Individuals with severe motion sickness or previous episodes of motion sickness due to VR (those who may not react well to the VR experience)
* Individuals with GFR<60 or previous documented diagnosis of CKD as they may not be suitable candidate for traditional analgesia
* Individuals with previous opioid dependence
* Requirement of immediate surgery (obstructing calculi with concomitant urinary tract infection)
* Patients with diagnoses meeting admission criteria (sepsis, MI)
* Audio/visual impairment (unable to appreciate stimuli provided by the headset)
* Patients administered opiates as the first line pain control medication will not be included in final data collection, as opioid administration may result in difficulty consenting and understanding the study protocol / design

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
60 Minute Pain Level | 60 minutes
  Pain Level Change 60 minutes after enrollment, utilizing a 0-10 subjective score

SECONDARY OUTCOMES:
30 Minute Pain Level | 30 minutes
  Pain Level 30 minutes after enrollment, utilizing a 0-10 subjective score
30 Minute Heart Rate | 30 minutes
  Change in Heart Rate 30 minutes after enrollment
30 Minute Blood Pressure | 30 minutes
  Systolic and Diastolic Blood Pressures 30 minutes after enrollment
60 Minute Heart Rate | 60 Minutes
  Change in Heart Rate 60 minutes after enrollment
60 Minute Blood Pressure | 60 minutes
  Systolic and Diastolic Blood Pressures 60 minutes after enrollment
Rescue Analgesia Use | 4 hours
  Requirement for Rescue Analgesia
Rescue Intervention | 24 Hours
  Requirement of Specialty Urologic Procedural Intervention for Pain Management (All Cause)

OTHER OUTCOMES:
Visual Analog Scale for Anxiety | 60 minutes
  Anxiety, as measured on a 10 cm line, with 0 being no anxiety, and 10 being worst anxiety patient has experienced, caused by AR Headset, to be measured in the AR Arm only
Subjective AR Experience | 60 minutes
  Likert Scale Response on if patient would use AR headset again, in AR arm only: 1 - Would Never Use Again; 2 - Would Consider Using Again; 3 - Neutral; 4 - Would Definitely Use Again if Offered; 5 - Would Ask to Use It Even if Not Offered

CONTACTS AND LOCATIONS:
Overall Officials: Chris Delmaestro, DO, Principal Investigator — Rutgers RWJBH Community Medical Center
Locations (1):
- Rutgers Robert Wood Johnson Barnabas Health Community Medical Center, Toms River, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weynants L, Chys B, D'hulst P, Merckx L, Van Besien J, Tailly T. Virtual reality for pain control during shock wave lithotripsy: a randomized controlled study. World J Urol. 2023 Feb;41(2):589-594. doi: 10.1007/s00345-023-04280-8. Epub 2023 Jan 21. PMID 36680576
- [Background] Pourmand A, Davis S, Marchak A, Whiteside T, Sikka N. Virtual Reality as a Clinical Tool for Pain Management. Curr Pain Headache Rep. 2018 Jun 15;22(8):53. doi: 10.1007/s11916-018-0708-2. PMID 29904806
- [Background] Mallari B, Spaeth EK, Goh H, Boyd BS. Virtual reality as an analgesic for acute and chronic pain in adults: a systematic review and meta-analysis. J Pain Res. 2019 Jul 3;12:2053-2085. doi: 10.2147/JPR.S200498. eCollection 2019. PMID 31308733
- [Background] Gottlieb M, Long B, Koyfman A. The evaluation and management of urolithiasis in the ED: A review of the literature. Am J Emerg Med. 2018 Apr;36(4):699-706. doi: 10.1016/j.ajem.2018.01.003. Epub 2018 Jan 5. PMID 29321112
- [Background] Holdgate A, Pollock T. Systematic review of the relative efficacy of non-steroidal anti-inflammatory drugs and opioids in the treatment of acute renal colic. BMJ. 2004 Jun 12;328(7453):1401. doi: 10.1136/bmj.38119.581991.55. Epub 2004 Jun 3. PMID 15178585
- [Background] Epidemiology of Nephrolithiasis. Course on Advances in Nephrology and Dialysis
- [Background] Worcester EM, Coe FL. Nephrolithiasis. Prim Care. 2008 Jun;35(2):369-91, vii. doi: 10.1016/j.pop.2008.01.005. PMID 18486720
- See also: Colorado Department of Public Health and Environment. Pain Scales. Colorado Department of Public Health and Environment, 2024 — https://cdphe.colorado.gov/sites/cdphe/files/OEPR5_CI_PainScales.pdf